CLINICAL TRIAL: NCT05379920
Title: Epigenetic and Cytokine Biomarkers During Recovery From Sports-Related Concussion
Brief Title: Salivary Biomarkers for Concussion Recovery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Praveen Arany, Associate Professor, State University of New York at Buffalo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00005734; UL1TR001412 (NIH)
Record Dates: First submitted 2022-03-01; First posted 2022-05-18 (Actual); Results first posted 2024-01-03 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Concussion, Brain
Keywords: adolescent; exercise; aerobic; biomarker; recovery
MeSH Terms: conditions — Brain Concussion; Motor Activity

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned into 4-arms: (1) Concussed participants: high volume exercise, (2) Concussed participants: low volume exercise, (3) Healthy controls: high volume exercise, (4) Healthy controls: low volume exercise. Each group will consist of 50% males and 50% females. Exercise interventions for all participants are adjusted to the 90% Heart rate threshold (HRt) collected on the BCTT. The high-volume group will exercise aerobically at 90% of their HRt for 5 days a week for 30 minutes. The low volume group will exercise aerobically at 90% of their HRt for 3 days a week for 30 minutes. The intervention will last 2 weeks. Participants will return to the clinic and repeat testing on Days 7 and 14. Recovery is defined as (1) resolution of concussion symptoms (2) physical examination within normal limits; (3) ability to exercise to at least 80% of age-appropriate maximum HR without exacerbation of concussion-like symptoms on the BCTT.
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Concussed Participants Group 1 (Experimental): High Volume Group
  Interventions: Behavioral: High Volume Aerobic Exercise
- Concussed Participants Group 2 (Experimental): Low Volume Group
  Interventions: Behavioral: Low Volume Aerobic Exercise
- Healthy controls Group 1 (Active Comparator): High Volume Group
  Interventions: Behavioral: High Volume Aerobic Exercise
- Healthy Controls Group 2 (Active Comparator): Low Volume Group
  Interventions: Behavioral: Low Volume Aerobic Exercise

INTERVENTIONS:
Behavioral: High Volume Aerobic Exercise — Aerobic exercise is completed for 30 minutes, 5 days a week. Exercise intensity is adjusted weekly to 90% of the heart rate threshold. Exercise interventions for all participants are adjusted to the 90% Heart rate threshold (HRt) collected on the BCTT.
  Arms: Concussed Participants Group 1; Healthy controls Group 1
Behavioral: Low Volume Aerobic Exercise — Aerobic exercise is completed for 20 minutes, 3 days a week. Exercise intensity is adjusted weekly to 90% of the heart rate threshold. Exercise interventions for all participants are adjusted to the 90% Heart rate threshold (HRt) collected on the BCTT.
  Arms: Concussed Participants Group 2; Healthy Controls Group 2

SUMMARY:
The overarching purpose of this proposed research is to determine whether BDNF and/or specific miRNAs can serve as biomarkers for recovery from a concussion during prescribed exercise. The investigators hypothesize salivary BDNF and specific miRNA signatures will change in a statistically significant manner as participants proceed from injury to recovery and participants who show recovery in ANS regulation will show significant differences in salivary BDNF and specific miRNA expression. This study also aims to determine if BDNF and/or specific miRNA can serve as biomarkers of the return of ANS function in concussed patients. The basic premise here is that the volume of exercise will significantly affect the rate of change in the expression of salivary BDNF and miRNA from injury to recovery.

DETAILED DESCRIPTION:
* This is a four-arm randomized control trial that investigates the changes in expression of BDNF/ miRNA after prescribed exercise intervention in concussed adolescents. Potential participants will be selected from incoming patients to the University Concussion Management Clinic. For a patient to become a potential participant in the "concussed participant" group, a sports medicine physician must first confirm the diagnosis of an acute concussion within 10 days of injury. Healthy controls will be recruited at local high schools (pediatric) and from the UB Clinical Trial registry (pediatric and adult). Concussion diagnosis is based on history, a concussion symptom questionnaire, and a concussion-specific physical examination. If the participant's medical history and demographic information meet eligibility criteria, they will be asked if they would like to participate. All potential participants will be informed of all study procedures verbally. If participants are willing and eligible to participate, they will be asked to consent/ assent to the study procedure.
* Participants will be asked to fill out the documentation regarding their demographics, concussion symptoms/history (Concussion Symptom Evaluation, Post-Concussion Symptom Inventory), and motivation to exercise (Modified Perceived Competence Scale, Modified Treatment Self-Regulation Questionnaire). Additionally, to determine if participants have any contraindications to exercise, the Physical Activity Readiness Questionnaire (PAR-Q) will be completed by all participants.
* Participants will undergo the Buffalo Concussion Physical Exam (BCPE), a short examination to used determine if a patient is concussed. This examination includes vital signs, a head and neck examination, cranial nerve testing, oculomotor testing, and a balance test.
* A trained examiner will complete an Oral Hygiene Index-Simplified (OHI-S) and will collect saliva. The Oral Hygiene Index is a short evaluation of the calculus and debris on selected teeth to assess the oral hygiene of a participant. Saliva will be collected using a Genotek Swab (miRNA) and a Salimetrics Cryovial (BDNF). Saliva will be collected with a swab (Genotek) and passive drool (Salimetrics) techniques.
* After saliva is obtained, the participant will be asked to complete the Buffalo Concussion Treadmill Test (BCTT). The BCTT is a graded exercise test that is used to determine concussion-related exercise intolerance. Although it is standard for patients from the Concussion Clinic to require a BCTT assessment as a part of their standard visit, participants will be made aware that their BCTT data will be used for this study. During the BCTT participants will be asked to wear an HR monitor (Polar H10) for the collection of HR and Heart Rate Variability (HRV) data.
* After completion of the BCTT, the examiner will use the results of the exercise test to create an individualized exercise prescription. The prescription will be randomized for high and low volumes and even split between male and female participants in healthy and concussed groups.
* Recovery date for concussed participants will be provided by the study clinician after the end of the intervention if concussed participants do not recover during the study time frame.

ELIGIBILITY:
Inclusion Criteria:

• Adolescent and adult athletes (age 13-18) diagnosed with SRC within 10 days of injury.

Exclusion Criteria:

* Evidence of focal neurological deficit;
* Inability to exercise because of orthopedic or cervical spine injury;
* Increased cardiac risk according to American College of Sports Medicine criteria;
* History of moderate or severe TBI, defined as brain injury with a Glasgow Coma Scale score of 12 or less;
* Current medication treatment for ADHD, learning disorders, depression, anxiety, or other medications that can affect HR;
* Symptom severity score of less than 5 on the initial visit Post Concussion Symptom Scale questionnaire. (7) currently pregnant (8) have any contraindications to exercise (Physical Activity Readiness-Questionnaire)

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Self-representation of gender identity
Enrollment: 60 (Actual)
Dates: Start 2022-03-22 (Actual); Primary Completion 2023-01-13 (Actual); Study Completion 2023-01-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Leddy, MD, Study Director — University at Buffalo; Barry Willer, PhD, Study Chair — University at Buffalo; Praveen Arany, DDS, PhD, Principal Investigator — University at Buffalo; Mohammad Nadir, MD, PhD, Study Director — University at Buffalo
Locations (1):
- UB MD Orthopeadics & Sports Medicine, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD currently

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited during the 1-year study beginning in 2022 from the UBMD Concussion Clinic. 32 concussed adolescents met inclusion criteria and were willing to participate in the study. Within the same time frame, 28 healthy adolescents were willing to participate in the study.
Period: Overall Study
Arm/Group | Concussed Participants Group 1 | Concussed Participants Group 2 | Healthy Controls Group 1 | Healthy Controls Group 2
Started | 17 | 15 | 15 | 13
Completed | 17 | 10 | 15 | 13
Not Completed | 0 | 5 | 0 | 0
Not completed — Lost to Follow-up | 0 | 5 | 0 | 0

BASELINE CHARACTERISTICS:
Population: It is hypothesized that participants in the concussion group would not different in age, sex, ethnicity, height or weight from control samples.
Groups:
- Total: Total of all reporting groups
Arm/Group | Concussed Participants Group 1 | Concussed Participants Group 2 | Healthy Controls Group 1 | Healthy Controls Group 2 | Total
Number analyzed (Participants) | 17 | 15 | 15 | 13 | 60
Age, Categorical [Count of Participants; unit: Participants] — Age Range in Years
  Participants
    <=18 years | 16 | 10 | 11 | 9 | 46
    Between 18 and 65 years | 1 | 5 | 4 | 4 | 14
    >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Binary sex as determined at birth
  Participants
    Female | 6 | 5. | 5 | 4 | 20
    Male | 11 | 10 | 10 | 9 | 40
Race (NIH/OMB) [Count of Participants; unit: Participants] — Racial ethnic group
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
    Asian | 0 | 0 | 1 | 1 | 2
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
    Black or African American | 0 | 2 | 1 | 1 | 4
    White | 15 | 12 | 13 | 9 | 49
    More than one race | 2 | 1 | 0 | 2 | 5
    Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants] — Geographical location of discrete groups
  participants
    United States | 17 | 15 | 15 | 13 | 60

OUTCOME MEASURES:

1. Primary Outcome: Persistent Post Concussion Symptoms (PPCS) (Yes/No)
Description: PPCS is defined as more recovery that occurs 28 days or more from the day of concussive injury (yes) or before 28 days (no). Recovery is defined as asymptomatic, exercise tolerant and confirmation by independent medical examination.
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Concussed Participants Group 1 | Concussed Participants Group 2
Number analyzed (Participants) | 17 | 15
Participants | 4 | 4

ADVERSE EVENTS:
Time Frame: Adverse events were monitored during the two week intervention.
Description: Adolescents participant condition (concussed or healthy) and intervention (light aerobic exercise) does not constitute a high risk for serious adverse events or mortality.
Arm/Group | Concussed Participants Group 1 | Concussed Participants Group 2 | Healthy Controls Group 1 | Healthy Controls Group 2
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/15 | 0/15 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/15 | 0/15 | 0/13
Other Adverse Events (participants affected / at risk) | 0/17 | 0/15 | 0/15 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-02): https://cdn.clinicaltrials.gov/large-docs/20/NCT05379920/Prot_SAP_000.pdf